CLINICAL TRIAL: NCT03037294
Title: Protein Turnover in the Osteoarthritic Knee; the Impact of Preoperative Protein Intake and Intra-articular Corticosteroid Injections
Brief Title: Protein Turnover in the Osteoarthritic Knee
Acronym: KneeT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Principal Investigator, Lex Verdijk, Assistant Professor, Maastricht University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 16-3-036
Record Dates: First submitted 2017-01-24; First posted 2017-01-31 (Estimated); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Osteo Arthritis Knee; Protein Metabolism

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (No Intervention): Subjects in the control group will receive no intervention.
- Protein group (Experimental): Subjects in the protein group will receive a daily 40 g pre-sleep protein supplement during the 2-week preoperative period.
  Interventions: Dietary Supplement: Preoperative protein supplementation

INTERVENTIONS:
Dietary Supplement: Preoperative protein supplementation — Daily 40 g of pre-sleep protein supplementation during 2-week preoperative period.
  Arms: Protein group

SUMMARY:
Rationale: Osteoarthritis (OA) of the knee is a common cause of pain and disability, especially in people over the age of 65. In the current health care system both conservative (e.g. intra-articular injections with corticosteroids) and surgical (total knee replacement, TKR) treatment are applied. Although frequently used, certain effects of these treatments on protein metabolism remain unclear. It is well known that maintenance of different tissues is determined by a dynamic balance between protein synthesis and breakdown rates, with temporary changes in either protein synthesis or breakdown allowing net protein accretion or loss. Though protein supplementation has shown to be an effective nutritional strategy in stimulating muscle protein synthesis, it remains unclear to what extent other musculoskeletal tissues are able to respond to dietary protein supplementation. Therefore, the current study assesses the impact of preoperative protein supplementation on protein synthesis in different musculoskeletal tissues of the knee.

Objective: To investigate the effect of preoperative protein supplementation on Hoffa's fat pad, synovium, tendon, bone, muscle, ligament, menisci, and cartilage protein synthesis of the OA knee.

Study design: Randomized, parallel (two groups) study design. The intervention group will be compared to the control group.

Study population: 24 adults with OA of the knee undergoing TKR. Intervention: Daily 40 g of pre-sleep protein two weeks before TKR or no intervention.

Main study parameters/endpoints: Primary study parameters include protein synthesis rates and enrichments of Hoffa's fat pad, synovium, tendon, bone, muscle, ligament, menisci, and cartilage. Secondary parameters include whole-body protein synthesis, breakdown, oxidation, and net balance.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: The risks involved in participating in this study are minimal. There are no potential effects known for the ingestion of protein. Muscle biopsies and tissue collection will be performed during the surgical procedure.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Male and female patients scheduled for total knee arthroplasty
* BMI between 18.5-30 kg/m2
* Age > 18 years
* Mentally competent, as judged by the treating physician
* Functioning gastrointestinal tract, eligible for oral protein supplementation

Exclusion Criteria:

* Corticosteroid injections less than 3 months prior to participation
* Any medications know to affect protein metabolism (i.e. corticosteroids, non-steroidal anti-inflammatories, or prescription strength acne medications)
* Lactose intolerance
* Insulin-dependent diabetes mellitus
* Alcohol abuse
* Rheumatoid arthritis
* Peripheral artery disease Fontaine III or IV
* COPD GOLD III or IV
* Phenylketonuria
* Surgical intervention in the past four weeks
* Total parenteral nutrition at day of surgery
* Neoadjuvant chemotherapy or radiotherapy
* GFR <20 mL/min/1.73 m2
* Osteoarthritis of the knee secondary to septic arthritis, osteonecrosis, fracture, OD, or malignant processes
* Collagen disorders, e.g. Marfan and Ehler-Danlos
* Any other medical condition that may interfere with the safety of the subjects or the outcome parameters, in the investigators judgement
* Investigator's uncertainty about the willingness or ability of the subject to comply with the protocol instructions
* Participation in any other studies involving investigational or marketed products concomitantly or within two weeks prior to entry into the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2024-01-19 (Actual); Study Completion 2024-01-19 (Actual)

PRIMARY OUTCOMES:
Change in tissue-specific protein synthesis rates | Throughout the surgical procedure (stable isotope methodology) and during the 2-week preoperative period (D2O dosing methodology).
  Fractional synthetic rates calculated based on tissue-free, plasma, and protein-bound tracer enrichments using stable isotope methodology and D2O dosing methodology.

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht University Medical Center, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: No